CLINICAL TRIAL: NCT05995652
Title: Can Shear Wave Elastography Predict the Success of Shock-Wave Lithotripsy Used in Renal Stones Treatment: a Prospective Study
Brief Title: Can Shear Wave Elastography Predict the Success of ESWL: a Prospective Study
Status: Completed | Type: Observational
Sponsor: Abdelrahim Elsherbiny (Other)
Responsible Party: Sponsor-Investigator, Abdelrahim Elsherbiny, assistant lecturer at urology department, Ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: Abdelrahim Elsherbiny
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESWL sucess and failed gps: post ESWL 50 pt large gp will be devided into sucess gp and failed gp
  Interventions: Procedure: elastography

INTERVENTIONS:
Procedure: elastography — elastography

SUMMARY:
Can Shear Wave Elastography predict the success of Shock-Wave Lithotripsy used in renal stones treatment ? A prospective study

DETAILED DESCRIPTION:
Extracorporeal shock-wave lithotripsy (ESWL) is the noninvasive treatment method that is recommended as the first choice in the treatment of small and medium sized renal stones and proximal ureteral stones.

This study is a trial to determine the predictive role of shear wave elastography in the success of ESWL management of kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years
* With single radiopaque renal stone
* Ranging in size from (1-1,5 cm) for ESWL.

Exclusion Criteria:

* Any urological abnormal anatomy
* Lower calyceal stone more than 1cm
* Impaired renal functions
* Uncorrected coagulopathy.
* Active UTI Pregnancy Single kidney Multiple stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1 gp of 50 pts will be subjected to ESWL and will be divided into 2 other gps success and failed
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
stone free rate | 1 month
  post ESWL

CONTACTS AND LOCATIONS:
Overall Officials: tarek elzayat, prof.dr., Study Chair — AinShams
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt